CLINICAL TRIAL: NCT01934478
Title: Study on Human Epidermal Growth Factor 2 (Her2) Expression Changes in Human Breast Cancer After Radiotherapy
Brief Title: Radiotherapy Alternates Human Epidermal Growth Factor 2 (Her2) Expression in Human Breast Cancer
Status: Completed | Type: Observational
Sponsor: Qingdao Central Hospital (Other)
Responsible Party: Principal Investigator, Youxin Ji, Chief, Department of Oncology, Qingdao Central Hospital
Other Study IDs: QCH20130823-2
Record Dates: First submitted 2013-08-23; First posted 2013-09-04 (Estimated); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Human Epidermal Growth Factor 2 Negative Carcinoma of Breast
Keywords: Breast; Cancer; Human Epidermal Growth Factor 2 (Her2); irradiation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Based on fundamental study （in Vitro and in Vivo, Pro. Jianjian Li）， Her2 expression would be changed from negative to positive by cancer irradiation with liner-accelerator at dose 6GY or up. The propose of this study is to reveal the irradiation result on Her2 expression in human breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* histological confirmed advanced breast cancer
* cancer sample can be obtained by fine needle biopsy
* IHC and FISH confirmed Her2 negative
* radiotherapy indication for local residual cancer

Exclusion Criteria:

* no radiotherapy indication
* patient refuse

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: study population is among advanced Chinese breast cancer patient.
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2013-08; Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Her2 changes during radiotherapy | every week up to 6 weeks
  biopsy is obtained by fine needle biopsy，Her2 is checked by Immunohistochemistry (IHC) and Fluorescence in situ hybridization (FISH).

CONTACTS AND LOCATIONS:
Overall Officials: ketao lan, M.D., Study Chair — Qingdao Health Bereau
Locations (1):
- Qingdao Central Hospital, Qingdao Cancer Hospital, Qingdao, Shandong, China